CLINICAL TRIAL: NCT03817736
Title: Sequential TransArterial Chemoembolization and Stereotactic RadioTherapy Followed by ImmunoTherapy for Downstaging Hepatocellular Carcinoma for Hepatectomy (START-FIT)
Brief Title: Sequential TACE and SBRT Followed by ImmunoTherapy for Downstaging HCC for Hepatectomy
Acronym: START-FIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Principal Investigator, Dr. Chi-Leung Chiang, Clinical Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 18-541
Record Dates: First submitted 2018-12-06; First posted 2019-01-25 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: HCC
Keywords: HCC; START-FIT; TACE; SBRT; immunotherapy; hepatectomy; hepatocellular carcinoma; liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- START-FIT (Experimental): Single group assignment combining TACE and SBRT with immune checkpoint inhibitor as treatment in HCC patients.
  Procedure of TACE will be standardized.
  SBRT screening and planning will be performed by radiation therapists, medical physicists, and oncologists.
  An immune checkpoint inhibitor may be administered up to 3 days before or after the scheduled day of administration of each cycle due to administrative reasons.
  Interventions: Procedure: TACE; Radiation: SBRT; Drug: Immune Checkpoint Inhibitor

INTERVENTIONS:
Procedure: TACE — Procedure of TACE will be standardized.
Radiation: SBRT — SBRT screening and planning will be performed by radiation therapists, medical physicists, and oncologists.
Drug: Immune Checkpoint Inhibitor — An immune checkpoint inhibitor may be administered up to 3 days before or after the scheduled day of administration of each cycle due to administrative reasons.

SUMMARY:
This study is a prospective phase II, single arm clinical study conducted in Queen Mary Hospital (Hong Kong) assessing the efficacy and safety of the sequential administration of trans-arterial chemo-embolization (TACE) and stereotactic body radiotherapy (SBRT) with an immune checkpoint inhibitor in hepatocellular carcinoma (HCC) patients.

DETAILED DESCRIPTION:
All the patients must be registered with the Investigator(s) prior to initiation of treatment. The registration desk will confirm all eligibility criteria and obtain essential information (including patient number).

TACE should start within 28 days of study registration and its procedure will be standardised.

SBRT screening and planning will be performed by radiation therapists, medical physicists, and oncologists.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of HCC confirmed pathologically or made according to American Association for the Study of Liver Diseases (AASLD) practice guideline 2010: patients with cirrhosis of any etiology and patients with chronic hepatitis B (HBV) who may not have fully developed cirrhosis, the presence of liver nodule >1cm and demonstrated in a single contrast-enhanced dynamic imaging [magnetic resonance imaging (MRI)] of intense arterial uptake and "washout" in portal venous and delayed phases.
2. Male or female subjects with age: 18-75 years old
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
4. Tumor size 5-15cm or number of lesions ≤3 or segmental portal vein involvement
5. Child-Pugh liver function class A-B7
6. Liver volume minus intrahepatic GTV >700 cc.
7. Minimal distance from GTV to stomach, duodenum, small or large bowel >1 cm.
8. No prior systemic therapy nor immunotherapy
9. No prior trans-arterial chemo-embolization (TACE)
10. No prior radiotherapy to the liver or selective internal radiation (SIRT)
11. Written informed consent obtained for clinical trial participation and providing archival tumor tissue, if available.
12. Subjects with confirmed concomitant HBV infection (defined as HBsAg positive or HBV DNA detectable) that are eligible for inclusion must be treated with antiviral therapy (per local institutional practice) prior to enrollment to ensure adequate viral suppression (HBV DNA <2000 IU/mL), must remain on antiviral therapy for the study duration, and continue therapy for 6 months after the last dose of investigational product(s)
13. At least one measurable lesion according to RECIST v1.1.
14. Adequate organ and marrow function, as defined below:

    * Hemoglobin ≥9 g/dL
    * Absolute neutrophil count ≥1,500/μL
    * Platelet count ≥100,000/μL
    * Total bilirubin ≤2.0 × ULN
    * ALT ≤3 × ULN
    * Albumin ≥2.8 g/dL
    * INR ≤1.6
    * Calculated creatinine clearance ≥45 mL/minute as determined by Cockcroft-Gault (using actual body weight) or 24-hour urine creatinine clearance
15. Females of childbearing potential or non-sterilized male who are sexually active must use a highly effective method of contraception
16. Females of childbearing potential must have negative serum or urine pregnancy test

Exclusion Criteria:

1. Prior invasive malignancy within 2 years except for noninvasive malignancies such as cervical carcinoma in situ, in situ prostate cancer, non-melanomatous carcinoma of the skin, lobular or ductal carcinoma in situ of the breast that has been surgically cured
2. Contraindicated of SBRT: Any one hepatocellular carcinoma >15 cm; Total maximal sum of hepatocellular carcinoma >20 cm; More than 3 discrete hepatic nodule; Direct tumor extension into the stomach, duodenum, small bowel, large bowel, common or main branch of biliary tree
3. Severe, active co-morbidity
4. Presence of extra-hepatic metastases (M1)
5. Left portal vein, right portal vein, main portal vein or inferior vena cava (IVC) thrombosis or involvement
6. Presence of clinically meaningful ascites as ascites requiring non pharmacologic intervention (eg, paracentesis) or escalation in pharmacologic intervention to maintain symptomatic control
7. Hepatic encephalopathy
8. Active or untreated gastrointestinal varices
9. Untreated central nervous system (CNS) metastatic disease, lepto-meningeal disease, or cord compression
10. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke ( <6 months prior to enrollment), myocardial infarction ( <6 months prior to enrollment), unstable angina, congestive heart failure (>= New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
11. Prior treatment with any immune checkpoint inhibitors or an antibody targeting immuno-regulatory receptors or mechanisms
12. Irritable bowel syndrome or other serious gastrointestinal chronic conditions associated with diarrhea within the past 3 years prior to the start of treatment
13. Known history of testing positive for HIV or known acquired immunodeficiency syndrome.
14. On chronic systemic steroid or any other forms of immunosuppressive medication within 14 days prior to the treatment. Except:

    1. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection);
    2. Systemic corticosteroids at physiologic doses <=10 mg/day of prednisone or equivalent;
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
15. Active or prior documented autoimmune or inflammatory disorders in the past 2 years, except diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment
16. History of primary immunodeficiency or solid organ transplantation
17. Receipt of live, attenuated vaccine within 28 days prior to the study treatment
18. Active infection requiring systemic therapy
19. Severe hypersensitivity reaction to treatment with another monoclonal antibody (mAb)
20. Females who are pregnant, lactating, or intend to become pregnant during their participation in the study
21. Psychiatric disorders and substance (drug/alcohol) abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Number of Patients Amendable to Curative Surgical Interventions | from the date of first study treatment to the date of last study treatment, an average of 3 years
  Number of patients amendable to curative surgical interventions defined as number of patients receiving curative surgical resection or transplantation after successful down-sizing of tumor(s) by intervention.

SECONDARY OUTCOMES:
Response rate measured by mRECIST criteria | from the date of screening to radiographically documented progression according to mRECIST 1.1, assessed up to 3 years
  Complete response (CR): Disappearance of any intra-tumoral arterial enhancement in all target lesions Partial response (PR): At least a 30% decrease in the sum of diameters of viable (enhancement in the arterial phase) target lesions, taking as reference the baseline sum of the diameters of target lesions Stable disease (SD): Any cases that do not qualify for either partial response or progressive disease Progressive disease (PD): An increase of at least 20% in the sum of the diameters of viable (enhancing) target lesions, taking as reference the smallest sum of the diameters of viable (enhancing) target lesions recorded since treatment started
Time to progression (TTP) | from the date of first study treatment to radiographically documented progression according to mRECIST 1.1, assessed up to 3 years
  Time to progression (TTP): measured from the date of first study treatment to radiographically documented progression according to mRECIST 1.1. This does not include death from any cause.
Progression-free survival (PFS) | from the date of first study treatment to radiographically documented progression according to mRECIST 1.1 or death from any cause, whichever occurs first, assessed up to 3 years
  Progression-free survival (PFS): measured from the date of first study treatment to radiographically documented progression according to mRECIST 1.1 or death from any cause (whichever occurs first). Participants alive and without disease progression or lost to follow-up will be censored at the date of their last radiographic assessment.
Overall survival (OS) | from the date of first study treatment to the date of death from any cause, assessed up to 5 years
  Overall survival (OS): measured from date of first study treatment to the date of death from any cause. Participants alive or lost to follow-up will be censored at the date of their last visit.
European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC-QLQ-C30) Score | from the date of screening to radiographically documented progression according to mRECIST 1.1, an average of 3 years
  Quality-of-Life (QoL) is assessed by the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC-QLQ-C30).
Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep) Score | from the date of screening to radiographically documented progression according to mRECIST 1.1, an average of 3 years
  Quality-of-Life (QoL) is also assessed by the Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep) questionnaires.
Incidence of Study-Related Adverse Events [Safety and Tolerability] | from the date of screening to 90 days after last treatment, around 3 years and 90 days
  Incidence, nature, and severity of adverse events graded according to the United States National Cancer Institute The Common Terminology Criteria for Adverse Events (NCI CTCAE 4.0)
Pathological response | from the date of first study treatment to radiographically documented progression according to mRECIST 1.1 or death from any cause, whichever occurs first, assessed up to 5 years
  Pathological response is assessed as the percentage of surface with non-viable cancer cells (represented by necrosis or fibrosis, the ultimate stage of necrosis) in relation to the total tumor area and will be equal to: 100% - viable cancer cells (%). If there are multiple tumors, the mean percentage will be used. Pathological complete response (pCR) is defined by the absence of viable tumor cells in any nodule.
Disease control rate | from the date of first study treatment to radiographically documented response according to mRECIST 1.1, assessed up to 3 years
  Percentage of patients that had a CR, PR, or SD ≥ 6 months per mRECIST
Local control | from the date of first study treatment to radiographically documented in-field progression according to mRECIST 1.1, censored at the time of intervention to target lesion, assessed up to 3 years
  Defined as absence of recurrence within the high-dose region (80% isodose volume), demonstrated by new enhancement or mRECIST progressive disease
Duration of response | from the date of first documented evidence of CR or PR to first documented sign of PD or death from any cause according to mRECIST 1.1, assessed up to 3 years
  Defined as the time from first documented evidence of CR or PR until the first documented sign of disease progression (PD) or death from any cause
Pattern of failure | from the date of first study treatment to radiographically documented failure type according to mRECIST 1.1, assessed up to 3 years
  (1) In-field failure: defined as recurrence within the high-dose region (80% iso-dose volume), demonstrated by new enhancement or mRECIST progressive disease; (2) Out-field (intra-hepatic): defined as new or mRECIST progressive disease within liver parenchyma, but outside the SBRT treated volume; (3) New vascular invasion: defined as new portal or hepatic vein invasion; (4) Distant failure: defined as new disease outside liver parenchyma

CONTACTS AND LOCATIONS:
Overall Officials: Chi Leung Chiang, Chiang, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Clinical Oncology, Hong Kong, Hong Kong

REFERENCES:
- [Background] Lo CM, Ngan H, Tso WK, Liu CL, Lam CM, Poon RT, Fan ST, Wong J. Randomized controlled trial of transarterial lipiodol chemoembolization for unresectable hepatocellular carcinoma. Hepatology. 2002 May;35(5):1164-71. doi: 10.1053/jhep.2002.33156. PMID 11981766
- [Background] Llovet JM, Real MI, Montana X, Planas R, Coll S, Aponte J, Ayuso C, Sala M, Muchart J, Sola R, Rodes J, Bruix J; Barcelona Liver Cancer Group. Arterial embolisation or chemoembolisation versus symptomatic treatment in patients with unresectable hepatocellular carcinoma: a randomised controlled trial. Lancet. 2002 May 18;359(9319):1734-9. doi: 10.1016/S0140-6736(02)08649-X. PMID 12049862
- [Background] Shim SJ, Seong J, Han KH, Chon CY, Suh CO, Lee JT. Local radiotherapy as a complement to incomplete transcatheter arterial chemoembolization in locally advanced hepatocellular carcinoma. Liver Int. 2005 Dec;25(6):1189-96. doi: 10.1111/j.1478-3231.2005.01170.x. PMID 16343071
- [Background] Llovet JM, Ricci S, Mazzaferro V, Hilgard P, Gane E, Blanc JF, de Oliveira AC, Santoro A, Raoul JL, Forner A, Schwartz M, Porta C, Zeuzem S, Bolondi L, Greten TF, Galle PR, Seitz JF, Borbath I, Haussinger D, Giannaris T, Shan M, Moscovici M, Voliotis D, Bruix J; SHARP Investigators Study Group. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med. 2008 Jul 24;359(4):378-90. doi: 10.1056/NEJMoa0708857. PMID 18650514
- [Background] Cheng AL, Kang YK, Chen Z, Tsao CJ, Qin S, Kim JS, Luo R, Feng J, Ye S, Yang TS, Xu J, Sun Y, Liang H, Liu J, Wang J, Tak WY, Pan H, Burock K, Zou J, Voliotis D, Guan Z. Efficacy and safety of sorafenib in patients in the Asia-Pacific region with advanced hepatocellular carcinoma: a phase III randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2009 Jan;10(1):25-34. doi: 10.1016/S1470-2045(08)70285-7. Epub 2008 Dec 16. PMID 19095497
- [Background] Blomgren H, Lax I, Naslund I, Svanstrom R. Stereotactic high dose fraction radiation therapy of extracranial tumors using an accelerator. Clinical experience of the first thirty-one patients. Acta Oncol. 1995;34(6):861-70. doi: 10.3109/02841869509127197. PMID 7576756
- [Background] Cardenes HR, Price TR, Perkins SM, Maluccio M, Kwo P, Breen TE, Henderson MA, Schefter TE, Tudor K, Deluca J, Johnstone PA. Phase I feasibility trial of stereotactic body radiation therapy for primary hepatocellular carcinoma. Clin Transl Oncol. 2010 Mar;12(3):218-25. doi: 10.1007/s12094-010-0492-x. PMID 20231127
- [Background] Andolino DL, Johnson CS, Maluccio M, Kwo P, Tector AJ, Zook J, Johnstone PA, Cardenes HR. Stereotactic body radiotherapy for primary hepatocellular carcinoma. Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):e447-53. doi: 10.1016/j.ijrobp.2011.04.011. Epub 2011 Jun 7. PMID 21645977
- [Background] Kang JK, Kim MS, Cho CK, Yang KM, Yoo HJ, Kim JH, Bae SH, Jung DH, Kim KB, Lee DH, Han CJ, Kim J, Park SC, Kim YH. Stereotactic body radiation therapy for inoperable hepatocellular carcinoma as a local salvage treatment after incomplete transarterial chemoembolization. Cancer. 2012 Nov 1;118(21):5424-31. doi: 10.1002/cncr.27533. Epub 2012 May 8. PMID 22570179
- [Background] Bujold A, Massey CA, Kim JJ, Brierley J, Cho C, Wong RK, Dinniwell RE, Kassam Z, Ringash J, Cummings B, Sykes J, Sherman M, Knox JJ, Dawson LA. Sequential phase I and II trials of stereotactic body radiotherapy for locally advanced hepatocellular carcinoma. J Clin Oncol. 2013 May 1;31(13):1631-9. doi: 10.1200/JCO.2012.44.1659. Epub 2013 Apr 1. PMID 23547075
- [Background] Radiation Therapy Oncology Group RTOG 1112 protocol. Available from: https://www.rtog.org/ClinicalTrials/ProtocolTable/StudyDetails.aspx?study=1112.
- [Background] Huo YR, Eslick GD. Transcatheter Arterial Chemoembolization Plus Radiotherapy Compared With Chemoembolization Alone for Hepatocellular Carcinoma: A Systematic Review and Meta-analysis. JAMA Oncol. 2015 Sep;1(6):756-65. doi: 10.1001/jamaoncol.2015.2189. PMID 26182200
- [Background] Hawkins MA, Dawson LA. Radiation therapy for hepatocellular carcinoma: from palliation to cure. Cancer. 2006 Apr 15;106(8):1653-63. doi: 10.1002/cncr.21811. PMID 16541431
- [Background] Chiang CL, Chan MKH, Yeung CSY, Ho CHM, Lee FAS, Lee VWY, Wong FCS, Blanck O. Combined stereotactic body radiotherapy and trans-arterial chemoembolization as initial treatment in BCLC stage B-C hepatocellular carcinoma. Strahlenther Onkol. 2019 Mar;195(3):254-264. doi: 10.1007/s00066-018-1391-2. Epub 2018 Nov 9. PMID 30413833
- [Background] Gehring AJ, Ho ZZ, Tan AT, Aung MO, Lee KH, Tan KC, Lim SG, Bertoletti A. Profile of tumor antigen-specific CD8 T cells in patients with hepatitis B virus-related hepatocellular carcinoma. Gastroenterology. 2009 Aug;137(2):682-90. doi: 10.1053/j.gastro.2009.04.045. Epub 2009 Apr 23. PMID 19394336
- [Background] Bernstein MB, Krishnan S, Hodge JW, Chang JY. Immunotherapy and stereotactic ablative radiotherapy (ISABR): a curative approach? Nat Rev Clin Oncol. 2016 Aug;13(8):516-24. doi: 10.1038/nrclinonc.2016.30. Epub 2016 Mar 8. PMID 26951040
- [Background] Postow MA, Callahan MK, Barker CA, Yamada Y, Yuan J, Kitano S, Mu Z, Rasalan T, Adamow M, Ritter E, Sedrak C, Jungbluth AA, Chua R, Yang AS, Roman RA, Rosner S, Benson B, Allison JP, Lesokhin AM, Gnjatic S, Wolchok JD. Immunologic correlates of the abscopal effect in a patient with melanoma. N Engl J Med. 2012 Mar 8;366(10):925-31. doi: 10.1056/NEJMoa1112824. PMID 22397654
- [Derived] Chiang CL, Chiu KWH, Chan KSK, Lee FAS, Li JCB, Wan CWS, Dai WC, Lam TC, Chen W, Wong NSM, Cheung ALY, Lee VWY, Lau VWH, El Helali A, Man K, Kong FMS, Lo CM, Chan AC. Sequential transarterial chemoembolisation and stereotactic body radiotherapy followed by immunotherapy as conversion therapy for patients with locally advanced, unresectable hepatocellular carcinoma (START-FIT): a single-arm, phase 2 trial. Lancet Gastroenterol Hepatol. 2023 Feb;8(2):169-178. doi: 10.1016/S2468-1253(22)00339-9. Epub 2022 Dec 15. PMID 36529152

DOCUMENTS (1):
  • Study Protocol (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/36/NCT03817736/Prot_002.pdf